CLINICAL TRIAL: NCT00970567
Title: Ketoacidosis in Individuals With T1DM
Brief Title: Ketoacidosis in Individuals With Type I Diabetes Mellitus (T1DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Abbott (Industry)
Responsible Party: Professor J. Spranger, Charité-Universitätsmedizin Berlin, Department of Endocrinology, Diabetes and Nutrition
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EA4/039/07
Record Dates: First submitted 2009-08-05; First posted 2009-09-02 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Type 1 Diabetes
Keywords: therapy after positive ketone bodies in the blood; timepoint of diagnosis; timepoint of metabolic normalisation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Other): stop after positive ketone bodies in urine
  Interventions: Behavioral: Different insulin therapy at different time points
- Arm 2 (Other): stop after positive ketone bodies in blood, normal therapy
  Interventions: Behavioral: Different insulin therapy at different time points
- Arm 3 (Other): stop after positive ketone bodies in blood, additional therapy
  Interventions: Behavioral: Different insulin therapy at different time points

INTERVENTIONS:
Behavioral: Different insulin therapy at different time points — different insulin therapy after positive blood ketones

SUMMARY:
The purpose of this study is to investigate individuals with type 1 diabetes who were disconnected from their insulin pump and insulin therapy was started again after positive ketones (U) in the urine or blood β-hydroxybutyrate.

DETAILED DESCRIPTION:
Individuals with type 1 diabetes were disconnected from their insulin pump and insulin therapy was started again after positive ketones (U) in the urine or blood β-hydroxybutyrate with different therapy regimens after positive blood ketones.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* severe hypo- or hyperglycemia during last 6 months
* acute illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
glucose metabolism, time course of positive ketone bodies | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Spranger, MD, Study Director — Charité, CBF
Locations (1):
- Charité-Universitätsmedizin Berlin, Department of Endocrinology, Diabetes and Nutrition, Berlin, State of Berlin, Germany